CLINICAL TRIAL: NCT03811262
Title: Comparison of Erector Spinae Plane Block With PECS II Block in Patients Undergoing Breast Cancer Surgery:a Randomized Controlled Trial
Brief Title: Comparison of Erector Spinae Plane Block With PECS II Block in Patients Undergoing Breast Cancer Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic reasons (Operating room performing the surgery investigated moved to another structure)
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESPvsPECS/AOP
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Anesthesia, Local
Keywords: PECS; ESP; RCT
MeSH Terms: conditions — Breast Neoplasms | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: This is a single-centre, prospective; double blinded randomised interventional clinical trial.
  Patients will be randomly allocated to group "PECS" or "ESP" using a closed envelope technique.
  Group "PECS" will receive PECS II block as described by Blanco using 30 ml Levobupivacaine 0.25% Group "ESP" will receive ESP block as described by forero using 30 ml Levobupivacaine 0.25% at T5 level.
  Blocks will be executed after general anesthesia induction. All partecipants will receive Fentanyl 2 mcg/kg and Propofol 2 mg/kg for induction. Anesthesia will be mantained with Propofol to obtain a BIS level between 40-50. Patients will receive Fentanyl 33 mcg whenever blood pressure and/or hear rate raise more than 20% from baseline after surgical stimulation. At the end of the surgery patients will receive acetominophen 1 g. postoperative therapy: acetominophen 1g/8hr and ketoprofen 100 mg/12hr.
  Patients will receive 2 mg Morphine whenever a NRS > 3.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: ESP block and PECS block will be executed by an anesthesiologist that will not follow the patient during the surgery.
  Anesthesiologist responsible for the surgery will be not aware of the block executed on the patient Anesthesiologist and surgeon responsible for postoperative therapy will be not aware of the block executed on the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP BLOCK (Active Comparator): Intervention:30 ml of 0.25% Levobupivacaine where: ESP block as described by Forero at T5 level (single injection between transversour process and erector spinae muscles)
  Interventions: Procedure: ESP BLOCK
- PECS block (Active Comparator): Intervention:30 ml of 0.25% Levobupivacaine where:PECS II block as described by Blanco.
  Interventions: Procedure: PECS BLOCK

INTERVENTIONS:
Procedure: ESP BLOCK — local anesthetic will be injected between transverous process and erector spinae muscle
  Arms: ESP BLOCK
Procedure: PECS BLOCK — local anesthetic will be injected between pectoralis minor and pectoralis major (10 ml) and between pectoralis minor and serratus (20 ml)
  Other Names: 30 ml 0.25% Levobupivacaine
  Arms: PECS block

SUMMARY:
Backgroung:Regional anesthesia in breast surgery is of paramount importance to reduce pain in perioperative period.

PECS II block is an interfascial block that has been used widely as regional anesthesia technique in breast surgery.

ESP block is a novel interfascial block proposed in 2016 by Forero. Several reports used this technique in breast surgery to provide analgesia but to date no studies comparing these technique exists.

Our hypotesis is that this two technique are equally able to provide analgesia in breast surgery.

Study type: RCT, single blind.

ELIGIBILITY:
Inclusion Criteria:

* Mastectomy program with axillary clearence

Exclusion Criteria:

* bilateral surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Fentanyl consumption | Intraoperative
  Intraoperative fentanyl dose (mcg) difference between ESP group and PECS group.

SECONDARY OUTCOMES:
NRS at 6 hour | sixth postoperative hour
  NRS (0-10) difference at sixth postoperative hour between ESP group and PECS group
NRS at 12 hour | twelth postoperative hour
  NRS (0-10) difference at twelth postoperative hour between ESP group and PECS group
NRS at 24 hour | twentyfourth postoperative hour
  NRS (0-10) difference at twentyfourth postoperative hour between ESP group and PECS group
Patient satisfaction at 24 hour | postoperative period (24h)
  Patient satisfaction (0-10) difference regarding anesthesia management at twentyfourth postoperative hour between ESP group and PECS group
Time to first opioid consumption in the postoperative period | postoperative period (24h)
  Time (minutes) to first opioid consumption in the postoperative period
Postoperative morphine consumption | postoperative period (24h)
  postoperative morphine dose (mg) difference between ESP group and PECS group.
Nausea and vomit incidence | postoperative period (24h)
  Incidence of nausea and vomiting in postoperative period
Other complication incidence | postoperative period (24h)
  Incidence of other complcations linked to anesthesia in postoperative period
Intraoperative Fentanyl consumption(mcg/kg/h) | Intraoperative
  Intraoperative fentanyl dose (mcg/kg/h) difference between ESP group and PECS group.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro De Cassai, MD, Principal Investigator — Department of Medicine, DIMED - Section of Anesthesiology and Intensive Care. University of Padova
Locations (1):
- University of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Probably data will be shared at the end of the study